CLINICAL TRIAL: NCT00503763
Title: Open -Label Phase IIa Trial of the Efficacy and Safety of Statin on the Course of Progressive Smoldering Multiple Myeloma
Brief Title: Efficacy and Safety of Statin on the Course of Progressive Smoldering Multiple Myeloma
Acronym: PSMMSS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We found out that there is another study on the same issue
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMMSS-01
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2007-07

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering multiple myeloma; Simvastatin; Paraprotein
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
The aim of the study is to evaluate the effect of statin administration on the course of progressive Smoldering Multiple Myeloma.

DETAILED DESCRIPTION:
In vitro data indicate that statins affect myeloma cells, mainly by inducing cell death and growth suppression.

This is a national, multicenter, phase IIa, single arm (not controlled), open label clinical trial of Simvastatin 80mg p.o. /day in a population of patients with progressive SMM. Patients will be treated with Simvastatin 40 mg and if no side effect will be seen the dose will be escalated to 80 mg for up to 18 months. All further treatment decisions after completion of the study are at the discretion of the investigator.Approximately 15 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling the criteria of SMM. (see Appendix I)
2. Patients with progressive smoldering Myeloma. (see Appendix II)
3. Age 18-80 years.
4. Signed informed consent prior to patient recruitment.

Exclusion Criteria:

1. Patients fulfilling diagnostic criteria of active MM .(see Appendix I)
2. Patients fulfilling diagnostic criteria of: solitary myeloma or non secreting myeloma or oligosecretory myeloma or light chain myeloma.
3. Patients on statin treatment on the day of recruitment.
4. Patients on chemotherapy or receiving steroids.
5. Patients with any contraindication to statin treatment:

   * Known intolerance or hypersensitivity to statin.
   * SGOT or SGPT above 1.5 times of upper normal level (UNL).
   * CPK above UNL
   * Concomitant treatment with macrolides and or antifungal agents (ketoconazole)
   * Creatinine level above 1.5 mg%
   * Any severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
6. Patients with second primary malignancy (except for non melanoma skin malignancy) unless they have been disease free for at least five years.
7. Patients who have a history of alcohol or drug abuse.
8. Patients who are mentally or physically unable to comply with all aspects of the study.
9. Participation to an investigational drug trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Paraprotein level | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lishner, MD, Principal Investigator — Meir Medical Center